CLINICAL TRIAL: NCT06551571
Title: The Effects of the Intrapartum Care Model Given in Line With the Recommendations of the World Health Organization (WHO) on the Mother's Maternal Behavior Towards Her Baby, Breastfeeding Self-efficacy, Breastfeeding Success, and Hospital Discharge Readiness
Brief Title: The Effects of the Intrapartum Care Model Given in Line With the Recommendations of the World Health Organization (WHO)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Seyhan Çankaya, Assoc. Prof. Seyhan Çankaya, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023/1143
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Birth Outcome, Adverse; Breast Feeding; Parenting
Keywords: WHO intrapartum care model; breastfeeding self-efficacy; LATCH; parenting behavior; discharge readiness
MeSH Terms: conditions — Pregnancy Complications; Breast Feeding

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): * In pregnant women with cervical dilatation of 5 cm, the Personal Information Form was completed at the initial clinic admission.
  * The Intrapartum Care Model was implemented for all primiparous pregnant women assigned to the intervention group during labor and after delivery by the researcher midwife, in accordance with the World Health Organization's positive birth recommendations.
  * The Postpartum Parenting Behavior Scale (PPBS), Breastfeeding Self-efficacy Scale (BSS), A Breastfeeding Charting System and Documentation Tool (LATCH), and Readiness for Hospital Discharge Scale-New Mother Form (RHD-NMF) were administered postpartum.
  Interventions: Other: Intrapartum Care Model
- Control Group (No Intervention): * Routine intrapartum care was provided to the pregnant woman in the hospital setting. This included taking an anamnesis, completing her file, opening an intravenous line, conducting routine blood tests, taking vital signs, recording cervical changes on the partograph via vaginal examination, applying EFM (electronic fetal monitoring) when indicated according to the attending physician's orders, listening to the fetal heart sounds (FHR) every fifteen minutes, and documenting this on the partograph.
  * The mother and infant received standard postpartum care in the hospital. Breastfeeding was initiated immediately after delivery, and the infant was placed in direct contact with the mother. The uterine tone and bleeding of the mother were evaluated, and vital signs were taken every four hours. Nutrition and mobilization were ensured, and a heel prick blood sample was taken in the 24th hour after delivery. If the mother and infant were normal after 24 hours, they were discharged.

INTERVENTIONS:
Other: Intrapartum Care Model — - The Intrapartum Care Model was implemented for all primiparous pregnant women assigned to the intervention group during labor and after delivery by the researcher midwife, in accordance with the World Health Organization's positive birth recommendations
  Arms: Intervention Group

SUMMARY:
The objective of this study was to examine the impact of the intrapartum care model that adheres to the guidelines set forth by the World Health Organization (WHO) on several key outcomes, including the mother's maternal behavior towards her infant postpartum, breastfeeding self-efficacy, the success of breastfeeding, and the mother's readiness for hospital discharge.

DETAILED DESCRIPTION:
The study was a randomized controlled trial. The study was conducted with 128 primiparous pregnant women (intervention group n=64, control group n=64) admitted to the maternity unit of a training and research hospital in a province in the Central Anatolia region of Turkey. Pregnant women in the intervention group were provided with intrapartum care in accordance with the WHO recommendations following the achievement of cervical dilatation reaching 5 cm. The control group was provided with only standard intrapartum and postpartum care. Data were collected using a personal information form, a postpartum parenting behavior scale, a breastfeeding self-efficacy scale, a breastfeeding charting system and documentation tool (LATCH), and a hospital discharge readiness scale.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older,
* History of term pregnancy (38-42 weeks),
* Having a primiparous,
* Single, healthy, vertex positioned fetus,
* Having no complications that may cause dystocia in labor (such as contraction anomalies, birth object,
* Birth canal dystocia, dystocia related to the mother's psychology),
* Having a partner/husband,
* History of cervical dilatation of 5 cm or more,
* Having a healthy newborn,
* Being able to speak and understand Turkish.

Exclusion Criteria:

* Being under 18 years of age,
* Having a diagnosed mental illness (depression, anxiety or other psychotic disorder, etc.),
* Having a chronic disease (hypertension, diabetes, etc.),
* Having maternal or fetal complications (oligohydramnios and polyhydramnios, placenta previa, pre-eclampsia, premature rupture of membranes, anomalies of presentation, intrauterine growth retardation, fetal anomaly, intrauterine death, fetal macrosomia, cord prolapse, etc.),
* Having any complication that prevents vaginal delivery (head-pelvis incompatibility, etc.),
* Having a history of elective cesarean section,
* Being pregnant with assisted reproductive techniques,
* Being multiparous,and having mastitis in the breast or having inverted nipples.
* The study also excluded women who had undergone a cesarean section due to any complication (e.g., cord entanglement, fetal distress),
* Who experienced complications related to the postpartum period (e.g., uterine atony, hemorrhage),
* And whose infant was admitted to the neonatal intensive care unit for any reason (e.g., respiratory distress).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Comparison of pre-intervention sociodemographic of pregnant women. | 6 months
  Sociodemographic of pregnant women will be collected through surveys and compared and reported
Comparison of pre-intervention obstetric features of pregnant women | 6 months
  Obstetric of pregnant women will be collected through surveys and compared and reported.
Comparison of postpartum characteristics of pregnant women | 6 months
  Postpartum characteristics of pregnant women will be collected through surveys and compared and reported.
Comparison of mother's postpartum parenting behavior towards her baby mean scores by groups | 6 months
  The postpartum parenting behavior scale will be applied to mothers. The postpartum parenting behavior scale is 0-6 points (min-max) and as the score increases, the level of positive parenting behaviors of mothers towards their babies increases.
Comparison of mother's breastfeeding self-efficacy scale mean scores by groups | 6 months
  The breastfeeding self-efficacy scale will be applied to mothers. The breastfeeding self-efficacy scale is 14-70 points (min-max) and as the score increases, the breastfeeding self-efficacy of the mothers increases.
Comparison of mother's A Breastfeeding Charting System and Documentation Tool (LATCH) mean scores by groups | 6 months
  The Breastfeeding Charting System and Documentation Tool (LATCH) will be applied to mothers.
  The LATCH is 0-10 points (min-max) and as the score increases, the LATCH of the mothers increases.
Comparison of mother's readiness for hospital discharge scale-new mother form mean scores by groups | 6 months
  The readiness for hospital discharge scale-new motherwill be applied to mothers.
  The readiness for hospital discharge scale-new mother is 0-220 points (min-max) and as the score increases shows that the mothers is sufficiently ready for discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Seyhan Çankaya, PhD, Principal Investigator — Selcuk University
Locations (1):
- Seyhan Çankaya, Konya, Turkey (Türkiye)